CLINICAL TRIAL: NCT04148339
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Elevated Cholesterol
Brief Title: A Pilot Study to Explore the Role of Gut Flora in Elevated Cholesterol
Status: Withdrawn | Type: Observational
Why Stopped: Company focus shifted
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-022
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cholesterol, Elevated; Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients with Elevated Cholesterol
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study.

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records regarding Elevated Cholesterol.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records regarding Elevated Cholesterol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
2. Male or female patients of any age (interest is given to children to compare with mothers).
3. LDL>100
4. Total Cholesterol>200

Exclusion Criteria:

1. Refusal to sign informed consent form
2. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
3. Postoperative stoma, ostomy, or ileoanal pouch
4. Participation in any experimental drug protocol within the past 12 weeks
5. Treatment with total parenteral nutrition
6. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
7. Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with elevated cholesterol
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Disease via Relative Abundance Found in Microbiome Sequencing | One year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific disease types.

SECONDARY OUTCOMES:
Validation of Sequencing Methods | One year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD